CLINICAL TRIAL: NCT00410813
Title: Phase II Studies of Two Different Schedules of Dasatinib (NSC-732517) in Bone Metastasis Predominant Metastatic Breast Cancer
Brief Title: S0622, Dasatinib in Treating Patients With Stage IV Breast Cancer That Has Spread to the Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000520348; S0622 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer; bone metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms, Male | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral dasatinib once daily.
  Interventions: Drug: dasatinib
- Arm II (Experimental): Patients receive oral dasatinib twice daily.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — given orally

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This randomized phase II trial is studying two different schedules of dasatinib to compare how well they work in treating patients with stage IV breast cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival of patients with stage IV bone metastasis-predominant breast cancer treated with 1 of 2 treatment schedules of dasatinib.
* Compare the response rate (complete and partial, confirmed and unconfirmed) in patients treated with these regimens.
* Compare the MUC-1 antigen response rate (CA 15-3 or CA 27-29) in patients treated with these regimens.
* Compare the circulating tumor cell response rate in patients treated with these regimens.
* Compare the anti-osteoclast activity, as measured by changes in bone turnover markers, in patients treated with these regimens.
* Compare the frequency and severity of toxicities of these regimens in these patients.
* Compare the pain profiles of these patients and explore changes over time.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to concurrent trastuzumab (Herceptin®) treatment (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dasatinib once daily.
* Arm II: Patients receive oral dasatinib twice daily. In both treatment arms, treatment continues for at least 24 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are acquired from patients once weekly in weeks 1, 4, 8, 16, and 24. Samples are analyzed for tumor markers, circulating tumor cells, and bone markers.

Patients complete a self-reported brief pain inventory questionnaire at baseline and once in weeks 8, 16, and 24.

After completion of study treatment, patients are followed every 3-6 months for up to 2 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast carcinoma meeting the following criteria:

  * Stage IV disease
  * Bone metastasis-predominant disease, defined as the presence of ≥ 1 bone metastasis with or without nonbone (visceral or soft tissue) disease where the number of bone metastases is at least the number of measurable visceral target lesions

    * Visceral disease that does not cause a reduction in ECOG performance status allowed
* Must meet 1 of the following criteria:

  * Measurable disease within the past 28 days
  * Nonmeasurable disease with rising serum CA 15-3, CA 27-29, CEA, or CA-125 documented by 2 consecutive measurements taken ≥ 14 days apart with the most recent measurement being within the past 42 days

    * These measurements need not be consecutive, and the prior measurement could have been months to years prior to the current measurement if the marker is considered by the investigator to reflect disease progression
    * The second serum marker value must be greater than the institution's upper limit of normal and show ≥ a 20% increase over the first measurement
* No symptomatic brain or CNS metastases

  * Prior CNS or brain metastasis allowed provided it was treated with radiotherapy ≥ 8 weeks ago
* No pleural or pericardial effusion
* Hormone receptor status known

  * Estrogen receptor- and/or progesterone receptor-positive disease must have progressed on ≥ 1 hormonal therapy in the metastatic setting

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Zubrod performance status 0-2
* QTc < 450 msec by EKG
* Ejection fraction ≥ 50% by MUGA or 2-dimensional echocardiogram with no significant abnormalities within the past 12 weeks for patients on trastuzumab
* No active infection requiring systemic therapy
* No uncontrolled concurrent condition that would preclude the ability to take oral medication, including the following:

  * Nausea
  * Vomiting
  * Diarrhea
  * Lack of physical integrity of the upper gastrointestinal tract
  * Malabsorption syndrome
* No clinically significant cardiac disease, including the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Cardiac arrhythmias not well controlled
  * Myocardial infarction within the past 12 months
* No concurrent active malignancy

  * Prior malignancies allowed provided the patient is currently disease-free
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior RankL inhibitor therapy
* No more than 1 prior cytotoxic chemotherapy for metastatic disease
* At least 3 weeks since prior chemotherapy and recovered
* At least 1 week since prior radiotherapy to non-CNS disease and recovered
* At least 3 weeks since prior and no concurrent intravenous bisphosphates (e.g., zoledronate)
* At least 7 days since prior and no concurrent antiplatelet agents, including any of the following*:

  * Anticoagulants (e.g., tirofiban, eptifibatide, ticlopidine)
  * Aspirin or aspirin-containing combinations
  * Dipyridamole
  * Epoprostenol
  * Clopidogrel
  * Cilostazol
  * Abciximab NOTE: *Nonsteroidal anti-inflammatory drugs and medically indicated platelet-inhibiting medication allowed
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * HIV protease inhibitors (e.g., amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir)
  * Select antibiotics (e.g., ciprofloxacin, clarithromycin, doxycycline, enoxacin, isoniazid, telithromycin)
  * Azole antifungals (e.g., itraconazole, ketoconazole, miconazole, voriconazole)
  * Select anesthetics (e.g., ketamine, propofol)
  * Hypericum perforatum (St. John's wort)
  * Nefazodone
  * Nicardipine
  * Diclofenac
  * Quinidine
  * Imatinib mesylate
* At least 7 days since prior and no concurrent medications that prolong the QTc interval, including any of the following:

  * Antiarrhythmic agents (e.g., quinidine, procainamide, disopyramide phosphate, amiodarone, sotalol hydrochloride, ibutilide, dofetilide)
  * Antipsychotic agents (e.g., chlorpromazine, mesoridazine, thioridazine, pimozide, haloperidol, droperidol)
  * Select antibiotics (e.g., erythromycin, clarithromycin, sparfloxacin, pentamidine)
  * Narcotic analgesics (e.g., levomethadyl, methadone, domperidone)
  * Calcium channel blockers (e.g., bepridil, lidoflazine)
  * Antimalarial agents (e.g., halofantrine, chloroquine)
  * Parasympathomimetic agents (e.g., cisapride)
  * Arsenic trioxide
* No other concurrent antineoplastic therapy for breast cancer, including any of the following:

  * Radiotherapy
  * Chemotherapy
  * Immunotherapy
  * Biologic therapy
  * Hormonal therapy
  * Gene therapy
* No concurrent grapefruit juice consumption
* No concurrent short-acting antacid agents within 2 hours of dasatinib administration
* Concurrent trastuzumab (Herceptin®) therapy for HER-2 positive patients allowed provided patients have been on continuous trastuzumab for ≥ 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-03; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne F. Schott, MD, Study Chair — University of Michigan Rogel Cancer Center; Catherine Van Poznak, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (117):
- United States (117):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Highlands Oncology Group - Springdale, Bentonville, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib, 100 mg, Daily: Dasatinib, 100 mg PO daily until progression of disease
- Dasatinib, 70 mg, Twice Daily: Dasatinib, 70 mg PO twice daily until progression of disease
Period: Overall Study
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Started | 43 | 42
Eligible | 41 | 38
Completed | 0 (Patients treated until progression.) | 0
Not Completed | 43 | 42
Not completed — Adverse Event | 6 | 11
Not completed — Progression | 32 | 21
Not completed — Not protocol specified | 3 | 4
Not completed — Ineligible | 2 | 4
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: All eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 82] | 65 [27 to 86] | 60 [27 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 38 | 35 | 73
  Black | 1 | 2 | 3
  Pacific Islander | 1 | 0 | 1
  Native American | 1 | 0 | 1
  Asian | 0 | 1 | 1
Use of trastuzumab at time of registration [Number; unit: participants]
  Yes | 1 | 0 | 1
  No | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: RECIST progression defined as 20% increase in the sum of longest diameters of target measurable lesions over the smallest sum observed, unequivocal progression of non-measurable disease, the appearance of any new lesion/site, death due to disease without prior documentation of progression and without symptomatic deterioration, development of one or more new bone lesions from baseline, or symptomatic deterioration related to disease progression. Time from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at last date of contact.
Time Frame: Up to 2 years
Population: All eligible patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 41 | 38
weeks | 10.3 [8.4 to 16.7] | 15.3 [8.7 to 20.1]

2. Secondary Outcome: Response Rate (Complete and Partial, Confirmed and Unconfirmed)
Description: Complete Response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions, no disease related symptoms, normalization of markers and other abnormal lab values. Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration. Progression is 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed, unequivocal progression of non-measurable disease, appearance of any new lesion/site, death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Up to 2 years
Population: All eligible patients
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 41 | 38
participants
  Partial Response | 1 | 0
  Stable/No Response | 14 | 18
  Increasing Disease | 20 | 10
  Assessment Inadequate | 6 | 10

3. Secondary Outcome: MUC-1 Antigen Response
Description: MUC-1 Complete Response is reduction in MUC-1 such that MUC-1 <= ULN. MUC-1 Partial Response is greater than or equal to a 50% reduction in MUC-1 from baseline, but not qualifying as a CR. MUC-1 Progression is greater than or equal to a 50% increase in MUC-1 from baseline. MUC-1 Stable Disease is MUC-1 response not qualifying as CR, PR, or Progression.
Time Frame: at 4, 8, 16, and 24 weeks
Population: MUC-1 Inadequate Assessment, response unknown: MUC-1 response has not been adequately assessed at indicated timepoints.
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Circulating Tumor Cells (CTC) Response Rate
Description: CTC response at 4 weeks is defined as the number of patients with initially elevated CTCs (>= 5 cells/7.5 ml), whose CTC level drops to < 5.
Time Frame: Up to 4 weeks
Population: Treatment arms are combined in this analysis. Only eligible patients evaluated at both baseline and at 4 weeks were included. Patients analyzed for CTC response only includes patients who had elevated CTCs at baseline.
Measure: Number; unit: participants
Groups:
- Dasatinib: Patients received either Arm 1: Dasatinib, 100 mg, daily or Arm 2: Dasatinib, 70 mg, twice daily.
Arm/Group | Dasatinib
Number analyzed (Participants) | 16
participants | 4

5. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time -- NTx
Description: Analysis included mean values of the serum biomarker NTx at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: nM BCE
Arm/Group | NTx at Baseline | NTx at 4 Weeks | NTx at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
nM BCE | 21.84 (12.32) | 19.23 (11.32) | 12.88 (13.09)

6. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time -- BAP
Description: Analysis included mean values of the serum biomarker BAP at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | BAP at Baseline | BAP at 4 Weeks | BAP at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
ug/L | 24.07 (15.95) | 24.35 (13.94) | 25.61 (14.05)

7. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time
Description: Analysis included mean values of the serum biomarkers sRANKL, IL-6, DKK, VEGF at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Serum Biomarker at Baseline | Serum Biomarker at 4 Weeks | Serum Biomarker at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
pg/mL
  DKK | 1157.64 (1465.83) | 1470.50 (1985.09) | 1575.05 (1993.44)
  IL-6 | 250.17 (1588.17) | 19.03 (73.70) | 32.03 (190.36)
  VEGF | 459.01 (324.89) | 424.21 (355.33) | 412.33 (346.58)
  sRANKL | 772172 (1580514) | 531173 (910765) | 553459 (864151)

8. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time -- OC
Description: Analysis included mean values of the serum biomarker OC at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OC at Baseline | OC at 4 Weeks | OC at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
ng/mL | 11.08 (7.76) | 13.10 (9.17) | 13.54 (10.20)

9. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time -- OPG
Description: Analysis included mean values of the serum biomarker OPG at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | OPG at Baseline | OPG at 4 Weeks | OPG at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
pmol/L | 4.56 (5.44) | 6.53 (9.46) | 6.71 (10.09)

10. Secondary Outcome: Change in Serum Bone Turnover Markers Over Time -- TRAP
Description: Analysis included mean values of the serum biomarker TRAP at baseline, 4, and 8 weeks.
Time Frame: at baseline, 4, and 8 weeks
Population: Number of patients with samples to analyze: baseline n=66, 4 weeks n=54, 8 weeks n=52.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | TRAP at Baseline | TRAP at 4 Weeks | TRAP at 8 Weeks
Number analyzed (Participants) | 66 | 54 | 52
U/L | 6.83 (6.42) | 5.41 (4.23) | 5.59 (4.40)

11. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 2 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE v3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 41 | 38
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 2
  AST, SGOT | 1 | 1
  Albumin, serum-low (hypoalbuminemia) | 0 | 1
  Anorexia | 0 | 1
  Dehydration | 0 | 1
  Diarrhea | 0 | 2
  Dyspnea (shortness of breath) | 1 | 4
  Fatigue (asthenia, lethargy, malaise) | 0 | 6
  Hemoglobin | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1 | 1
  Infection with unknown ANC - Dental-tooth | 1 | 0
  Left ventricular systolic dysfunction | 2 | 1
  Lymphopenia | 0 | 1
  Nausea | 0 | 1
  Neutrophils/granulocytes (ANC/AGC) | 0 | 1
  Pain - Bone | 1 | 1
  Pain - Buttock | 1 | 0
  Pain - Chest wall | 1 | 0
  Pain - Chest/thorax NOS | 1 | 0
  Pain - Head/headache | 1 | 1
  Platelets | 2 | 1
  Pleural effusion (non-malignant) | 1 | 2
  Pneumonitis/pulmonary infiltrates | 1 | 0
  Potassium, serum-low (hypokalemia) | 1 | 3
  Pulmonary hypertension | 0 | 1
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1
  Rash/desquamation | 0 | 1
  Sodium, serum-low (hyponatremia) | 0 | 1
  Vomiting | 0 | 1

12. Secondary Outcome: Mean Patient-reported Pain
Description: Patient's rating of "worst pain" experienced between prestudy and week 24. Changes of >=2 points on the Brief Pain Inventory (BPI) are of interest. Pain is self-reported on the Brief Pain Inventory Short Form, on a 0-10 response scale, with higher scores reflecting more pain and more interference with functioning.
Time Frame: Baseline, 8, 16, and 24 weeks
Population: All patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dasatinib - Baseline; Dasatinib - Week 8; Dasatinib - Week 16; Dasatinib - Week 24: Patients received either Arm 1: Dasatinib, 100 mg, daily or Arm 2: Dasatinib, 70 mg, twice daily.
Arm/Group | Dasatinib - Baseline | Dasatinib - Week 8 | Dasatinib - Week 16 | Dasatinib - Week 24
Number analyzed (Participants) | 79 | 68 | 37 | 41
units on a scale | 3.37 (2.93) | 3.82 (3.04) | 3.06 (2.61) | 3.73 (3.03)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Dasatinib, 100 mg, Daily | Dasatinib, 70 mg, Twice Daily
Serious Adverse Events (participants affected / at risk) | 6/41 | 12/38
Other Adverse Events (participants affected / at risk) | 34/41 | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg, Daily (N=41) | Dasatinib, 70 mg, Twice Daily (N=38)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1 | 1
Rash: dermatitis associated w/Chemoradiation (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg, Daily (N=41) | Dasatinib, 70 mg, Twice Daily (N=38)
Hemoglobin (Blood and lymphatic system disorders) | 16 | 22
Constipation (Gastrointestinal disorders) | 8 | 3
Diarrhea (Gastrointestinal disorders) | 10 | 14
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 3 | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 15 | 19
Vomiting (Gastrointestinal disorders) | 10 | 8
Edema: head and neck (General disorders) | 1 | 3
Edema: limb (General disorders) | 2 | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 | 19
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3 | 2
Pain - Chest/thorax NOS (General disorders) | 2 | 2
Pain-Other (Specify) (General disorders) | 5 | 5
Rigors/chills (General disorders) | 1 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 3 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 | 12
AST, SGOT (Investigations) | 10 | 16
Alkaline phosphatase (Investigations) | 6 | 9
Creatinine (Investigations) | 5 | 6
Leukocytes (total WBC) (Investigations) | 7 | 7
Lymphopenia (Investigations) | 2 | 3
Metabolic/Laboratory-Other (Specify) (Investigations) | 0 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 | 4
Platelets (Investigations) | 4 | 5
Weight loss (Investigations) | 2 | 6
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 6
Anorexia (Metabolism and nutrition disorders) | 8 | 9
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11 | 9
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 | 9
Pain - Back (Musculoskeletal and connective tissue disorders) | 12 | 4
Pain - Bone (Musculoskeletal and connective tissue disorders) | 7 | 10
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 4 | 1
Neuropathy: sensory (Nervous system disorders) | 6 | 3
Pain - Head/headache (Nervous system disorders) | 11 | 9
Taste alteration (dysgeusia) (Nervous system disorders) | 2 | 4
Tremor (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 7 | 4
Mood alteration - anxiety (Psychiatric disorders) | 6 | 4
Mood alteration - depression (Psychiatric disorders) | 3 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 2
Urine color change (Renal and urinary disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 | 6
Hot flashes/flushes (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less